CLINICAL TRIAL: NCT07183345
Title: Application of Dynamic Pain Assessment and Management System in Perioperative Period of Patients With Incarcerated Mixed Hemorrhoids: A Single-Center, Prospective, Open-Label, Randomized Controlled Trial
Brief Title: Application of Dynamic Pain Assessment and Management System in Perioperative Period of Patients With Incarcerated Mixed Hemorrhoids
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: putianU-006
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Incarcerated Mixed Hemorrhoids
Keywords: Pain Management; Preoperative Analgesia; Traditional Chinese Medicine (TCM) Fumigation; Wrist-Ankle Acupuncture (WAA); Dynamic Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): adopted routine drug analgesia
  Interventions: Drug: Routine drug analgesia
- study group (Other): Adoption of a Dynamic Pain Assessment and Management System
  Interventions: Other: Dynamic Pain Assessment and Management System

INTERVENTIONS:
Other: Dynamic Pain Assessment and Management System — Personalized nursing education was adopted. These measures include the use of preoperative analgesic drugs, postoperative Traditional Chinese Medicine (TCM) fumigation, and wrist-ankle acupuncture for pain relief.
  Arms: study group
Drug: Routine drug analgesia — adopted routine drug analgesia and conventional nursing education
  Arms: control group

SUMMARY:
This study aims to investigate whether the dynamic pain assessment and management system can alleviate postoperative pain in patients with incarcerated mixed hemorrhoids and reduce the incidence of complications. A total of 64 eligible patients were enrolled and randomly divided into two groups, with the specific grouping and intervention methods as follows:

① Control Group: Routine drug analgesia and conventional nursing education were adopted.

② Study Group: Patients were managed with the dynamic pain assessment and management system, which included preoperative administration of analgesic drugs, postoperative traditional Chinese medicine (TCM) fumigation, wrist-ankle acupuncture for pain relief, and personalized nursing education.

The study evaluated the effect of the dynamic pain assessment and management system on postoperative analgesia by comparing the Numerical Rating Scale (NRS) scores for pain, recording the Visual Analogue Scale (VAS) scores for quality of life, and analyzing the incidence of complications among patients in different groups. The primary hypothesis of the study is that, compared with routine pain management methods, the dynamic pain assessment and management system can significantly reduce postoperative pain in patients, improve their quality of life, and decrease the incidence of complications (such as bleeding and urinary retention).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years old
* Diagnosed with grade III-IV incarcerated mixed hemorrhoids according to the Goligher classification
* Undergoing standard hemorrhoidectomy
* Receiving simple intraspinal anesthesia

Exclusion Criteria:

* Pregnant or lactating patients
* Patients receiving immunotherapy or with coagulation dysfunction
* Patients who need to use various analgesic drugs daily
* Complicated with other anorectal diseases (such as perianal abscess, anal fistula, anal incontinence)
* Complicated with other systemic diseases (cardiac insufficiency; hepatic or renal insufficiency; diabetes mellitus; coagulation disorders; peptic ulcer, etc.)
* Incomplete perioperative clinical data
* Unable to cooperate with follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale (NRS) | Baseline, Day 1, 3, 5, 7, and Day 14±2
  The NRS uses a linear numerical range of "0 to 10" to represent pain intensity. Patients select the corresponding number based on their own perception, where a score of 0 indicates no pain at all, and a score of 10 represents the most severe pain you can imagine.

SECONDARY OUTCOMES:
Incidence Rate of Complications | within 30 days after surgery
  Measurements include the incidence rate of complications such as postoperative hemorrhage and urinary retention
Length of Hospital Stay | from the end of surgery to discharge (a maximum of 7 days)
  with hours as the unit, and standardized discharge criteria are adopted.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, China

IPD SHARING:
Plan to Share IPD: No
Based on a strict commitment to participant privacy protection, compliance with the terms of the ethical review protocol, and adherence to the sponsoring institution's policies, IPD from this study will not be shared at this time.